CLINICAL TRIAL: NCT04381507
Title: CONFORM-TAA - a Post-market Clinical Follow-up Study in Patients with a Descending Thoracic Aortic Aneurysm or Penetrating Aortic Ulcer (PAU) Treated with the E-nya Thoracic Stent Graft System
Brief Title: A Study in Patients with a Descending TAA or PAU Treated with the E-nya Thoracic Stent Graft System
Acronym: CONFORM-TAA
Status: Terminated | Type: Observational
Why Stopped: Expiry of CE mark.
Sponsor: JOTEC GmbH (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Other Study IDs: CONFORM-TAA
Record Dates: First submitted 2020-05-02; First posted 2020-05-11 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Vascular Aneurysm
Keywords: Descending; Aorta; Penetrating; Ulcer
MeSH Terms: conditions — Ulcer | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: endovascular repair — Endovascular repair of descending thoracic aneurysms or PAU using a stent graft.

SUMMARY:
The CONFORM-TAA post-market clinical follow-up study is undertaken to evaluate the prevention of death related to a descending aortic aneurysm or PAU when treated by the E-nya Thoracic Stent Graft System. The secondary objective is to evaluate the safety and clinical performance of the device.

DETAILED DESCRIPTION:
In this study, patients who receive an E-nya Thoracic Stent Graft for the endovascular treatment of descending thoracic aortic aneurysm or PAU will be observed. The E-nya Thoracic Stent Graft will be implanted in accordance with the instructions for use of the E-nya Thoracic Stent Graft System and at the discretion of the treating physician.

Participating physicians will be asked to provide their observations collected during routine standard of care for patients he/she had decided to treat with the E-nya Thoracic Stent Graft System. Informed consent of the patients will be obtained to allow the use of their clinical records for the purpose of this observational study before data are being collected.

The period of data collection for each patient will be approximately 60 months from the intervention. Source document verification will be performed on 100% of patients; data from all visits will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans will be sent to the CoreLab for independent evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* A fusiform focal TAA ≥ 55 mm for females, ≥ 60 mm for males, or ≥ 2 times the diameter of the non-aneurysmal thoracic aorta and/or focal saccular TAA or penetrating aortic ulcer (PAU)
* Suitable proximal and distal landing zone in the native aorta
* Landing zone of the proximal edge of the fabric distal to the left carotid artery
* Landing zone of the distal edge of the fabric proximal to the celiac trunk
* Proximal and distal non-aneurysmal neck diameter between 18 and 42 mm
* Proximal non-aneurysmal neck length ≥ 20 mm
* Distal non-aneurysmal neck length ≥ 20 mm
* Thoracic aortic lesion confirmed by thin sliced (≤ 1 mm) CTA with optional three-dimensional reconstruction obtained within 3 months prior to the implant procedure
* Patient is able and willing to undergo follow-up imaging and examinations prior to discharge from the hospital, at 30 days and 12 months, and annually thereafter until 5 years follow-up
* Patient understands and has signed the Informed Consent Form prior to intervention

Exclusion Criteria:

* Female of child bearing potential, breast feeding
* Access vessels not suitable for endovascular treatment
* Significant circular thrombi or calcification in proximal or distal landing zones
* Genetic connective tissue diseases (e.g. Marfan syndrome or Ehler-Danlos Syndrome)
* Allergies against materials necessary for endovascular repair (e.g. contrast media, heparin, materials of the stent graft)
* Systemic or local infections
* eGFR < 45 ml/min/1.73m2 before the intervention
* Mycotic aneurysm
* Myocardial infarction or cerebrovascular accident < 3 months ago
* Patient has specified disease of the thoracic aorta which is not included in the registry, for example: aortic dissection, intramural hematoma, traumatic injury or transection, aortic false aneurysm, (contained) ruptured aneurysm
* Patients who are planned to be treated with a chimney in the left subclavian artery
* Treatment of a thoracoabdominal or infrarenal aneurysm at the time of implant
* Previous stent and/or stent graft or previous surgical repair of descending thoracic aorta
* Patient had or planned to have a major surgical or interventional procedure within 30 days before or 30 days after the planned implantation of the E-nya Stent Graft System(s). This exclusion does not include planned procedures that are needed for the safe and effective placement of the stent graft (ie, carotid/subclavian transposition, carotid/subclavian bypass procedure)
* Other medical condition that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with a limited life expectancy (i.e. heart failure, active malignancy (progressive, stable or partial remission))
* Simultaneously participating in another clinical trial
* NYHA class IV

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with descending thoracic aortic aneurysm or PAU and who are eligible for treatment with a thoracic stent graft according to the instructions for use for the E-nya Thoracic Stent Graft System and scheduled for implantation of the E-nya Thoracic Stent Graft System at their physician's discretion in accordance with the listed inclusion / exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of all-cause mortality during the peri-operative period
Mortality | 12, 24, 36, 60 months
  Rate of all-cause mortality
Mortality | 30-day, 12, 24, 36, 60 months
  Rate of aneurysm / PAU related mortality
Rupture | 30-day, 12, 24, 36, 60 months
  Rate of patients with aneurysm / PAU rupture
Primary technical success | 24 hours
  Primary technical success related to the E-nya Thoracic Stent Graft System combines the following criteria:
  * It is related to periprocedural events that occur from the initiation of the procedure and extend through the first 24-hours postoperative period
  * Defined on an intent-to-treat basis
  * Successful access to the arterial system using a remote site (ie, the femoral, external iliac, common iliac, abdominal aorta, or brachiocephalic arteries with or without use of a temporary or permanent prosthetic conduit to access these arteries)
  * Successful deployment of the endoluminal graft at the intended location
  * Absence of reintervention, surgical conversion to open repair or death ≤24 h
Technical success | 24 hours
  Technical success is achieved in case all above mentioned criteria are fulfilled however, a reintervention was performed.
Primary clinical success | prior to discharge/30-day, 12, 24, 36, and 60 months
  Primary clinical success related to the E-nya Thoracic Stent Graft combines the following criteria:
  * Clinical success should be reported on an intent-to-treat basis
  * Initially required successful deployment of the E-nya Thoracic Stent Graft at the intended location without any
    * Death as a result of the pathology that was treated
    * Rupture of descending thoracic aortic aneurysm or PAU
    * Conversion to open repair
    * Reintervention
    * E-nya Thoracic Stent Graft infection
    * E-nya Thoracic Stent Graft infolding
    * Causing a new thoracic aortic pathology as a result of the intervention (eg, pseudoaneurysm, dissection, intramural hematoma, fistula)
Clinical success | prior to discharge/30-day, 12, 24, 36, and 60 months
  Clinical success is achieved in case all above mentioned criteria are fulfilled however, a reintervention was performed.
Major adverse event(s) | 30-day, 12, 24, 36, and 60 months
  Rate of patients with major adverse event(s) (death, aneurysm rupture, conversion to open surgical repair, retrograde type A dissection, stent graft induced postimplantation dissection requiring intervention, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke, new permanent paraplegia, new permanent paraparesis, new chronic renal insufficiency/renal failure requiring dialysis, bowel resection, > 72 hours artificial respiratory assistance, device induced trauma requiring intervention) (product related, procedure related, aneurysm related)
Conversion to open surgery | 24hours, 30-day, 12, 24, 36, and 60 months
  Rate of patients with conversion to open surgical repair
Reintervention | 30-day, 12, 24, 36, and 60 months
  Rate of patients with reintervention(s)
Aneurysm size | 12, 24, 36, and 60 months
  Rate of patients with decreasing (<5 mm), stable, increasing (>5 mm) aneurysm size
Endoleak Type Ia | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with type Ia endoleak
Endoleak Type Ib | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with type Ib endoleak
Endoleak Type II | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with type II endoleak
Endoleak Type III | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with type III endoleak
Endoleak Type IV | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with type IV endoleak
Cerebrovascular event | 30-day, 12, 24, 36, and 60 months
  Rate of patients with new cerebrovascular event/stroke (excluding transient ischemic attack)
Permanent paraplegia | 30-day, 12, 24, 36, and 60 months
  Rate of patients with new new permanent paraplegia
Permanent paraparesis | 30-day, 12, 24, 36, and 60 months
  Rate of patients with new new permanent paraparesis
Migration | prior to discharge/30-day, 12, 24, 36, and 60 months
  • Rate of E-nya Stent Graft migration:
  * Rate of patients with proximal E-nya Stent Graft migration (>5 mm)
  * Rate of patients with distal E-nya Stent Graft migration (>5 mm)
Dislodgement | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with E-nya Stent Graft dislodgement (full component separation)
Integrity | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with failure of E-nya Stent Graft integrity (stent fracture, fabric erosion)
Infolding | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with infolding of an E-nya Stent Graft

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brunkwall, Prof., Study Director — Brumed; Jost P. Schäfer, Prof., Study Chair — University Hospital Schleswig-Holstein (UKSH) Kiel
Locations (1):
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany